CLINICAL TRIAL: NCT05658380
Title: Impact of Pre-spinal Atropine on Post Spinal Hemodynamics and Cardiac Output Measured by Electrical Cardiometry in Caesarean Delivery: Randomized Double Blinded Controlled Trial
Brief Title: Impact of Pre-spinal Atropine on Post Spinal Hemodynamics and Cardiac Output Measured by Electrical Cardiometry in Caesarean Delivery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amin Mohammed Alansary Amin Ahmed Helwa, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R216/2022
Record Dates: First submitted 2022-12-04; First posted 2022-12-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Anesthesia
MeSH Terms: interventions — Atropine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- atropine (Active Comparator)
  Interventions: Drug: atropine
- normal saline (Placebo Comparator)
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: atropine — patients will receive 0.01 mg/kg intravenous atropine in 5 ml normal saline 0.9 % before induction of spinal anaesthesia
  Arms: atropine
Drug: Isotonic saline — patients will receive the same volume of isotonic saline 0.9% 5ml (control group) before induction of spinal anaesthesia
  Arms: normal saline

SUMMARY:
Cesarean section is one of the most commonly performed surgical procedures; approximately 80-90% of elective cesarean sections are conducted using spinal anesthesia . Spinal anesthesia is the preferred technique for Cesarean Section (CS) due to its simplicity, reliability, low rates of airway complications, facilitation of postoperative analgesia, less neonatal exposure to potentially depressant drugs, to awake mother at the time of the birth of the child that establishes maternal-infant bonding and successful breastfeeding, and due to its low cost as compared to the general anesthesia . The chance of significant maternal hypotension is greater with spinal anesthesia than with epidural anesthesia. Left uterine displacement with appropriate administration of fluids and use of vasopressor medications can minimize the associated hypotension. Intravenous administration of crystalloid or colloid can reduce the degree of hypotension after spinal anesthesia for cesarean delivery.

Maternal hypotension is a frequent side effect of spinal anesthesia for cesarean delivery and it causes dangerous maternal and fetal effects . Maternal hypotension decreases uteroplacental circulation and it results in nausea, vomiting, bradycardia and different systems dysfunction particularly in the presence of other diseases as renal, hepatic, cardiac and neurological. Anesthesiologists should not allow hypotension to continue, this often requires the use of vasopressors to maintain blood pressure as ephedrine, phenylephrine and norepinephrine .

Cardiac output is the amount of blood pumped by the heart per unit of time and is determined by four factors: two factors that are intrinsic to the heart-heart rate and myocardial contractility-and two factors that are extrinsic to the heart -preload and afterload. Heart rate is defined as the number of beats per minute and is mainly influenced by the autonomic nervous system. Increases in heart rate escalate cardiac output if ventricular filling is adequate during diastole .

Atropine is an anticholinergic agent with its ability to treat bradycardia both in mother and fetus. Atropine is an anti-sialagogue as well as used to antagonize the muscarinic side effects of anticholinesterases. Atropine is detected in the umbilical circulation within 1 to 2 minutes of maternal administration, and an F/M ratio of 0.93 is attained at 5 minutes .

ELIGIBILITY:
Inclusion Criteria:

* American society of anaesthesiologists (ASA) II
* full term
* singleton
* pregnant women scheduled for elective Cs

Exclusion Criteria:

* patients refusal
* with body mass index (BMI) > 35 Kg/m2
* polyhydramnios
* history of impaired cardiac contractility
* valvular heart disease
* cardiac arrhythmias
* hypertensive pregnancy disorders
* thyrotoxicosis
* cerebrovascular diseases
* foetal abnormalities
* Contraindications to spinal anesthesia as coagulopathy, infection at the site of needle insertion
* uncorrected hypovolemic shock
* increased intracranial pressure from mass effect
* inadequate resources or expertise.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-25 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
change in cardiac output measurment | basline and 5 minute after spinal anesthesia
  change in cardiac output (CO) will be measured by electrical cardiometry

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt